CLINICAL TRIAL: NCT01714414
Title: A Prospective, Multicenter, Open, Randomized Phase 2a Trial to Confirm a Sustained Virological Suppression Defined as HIV-RNA <50 Copies/ml of 3 Different Doses of Fozivudine in Context to a Standard Zidovudine Based Antiretroviral Therapy Regimen After 24 Weeks of Treatment in ART naïve, Non Subtype B HIV-1 Infected Individuals From Tanzania and Ivory Coast
Brief Title: A Trial to Confirm a Sustained Virological Suppression Defined as HIV-RNA <50 Copies/ml of 3 Different Doses of Fozivudine in Context to a Standard Zidovudine Based Antiretroviral Therapy Regimen
Acronym: FATI-01
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Michael Hoelscher (Other)
Collaborators: European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government); German Federal Ministry of Education and Research (Other Government); National Institute for Medical Research, Tanzania (Other Government); Treichville Academic hospital center, Division of infectious and tropical diseases (SMIT) (Unknown); ANRS, Emerging Infectious Diseases (Other Government); Kumasi Centre for Collaborative Research (KCCR) (Other); Bernhard Nocht Institute for Tropical Medicine (Other Government); Pharmaceutical Company (Chiracon GmbH) (Unknown); Pharmaceutical Company (STADA Vietnam Joint Venture Co. Ltd.) (Unknown)
Responsible Party: Sponsor-Investigator, Michael Hoelscher, Chief Investigator, Ludwig-Maximilians - University of Munich
Organization: Ludwig-Maximilians - University of Munich (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LMU-IMPH-FATI-01
Record Dates: First submitted 2012-10-25; First posted 2012-10-26 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: HIV-1 Infection
Keywords: HIV; Fozivudine; Zidovudine; FATI
MeSH Terms: interventions — fozivudine tidoxil; Lamivudine; efavirenz; Zidovudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- FZD 600mg twice daily (Experimental): FZD 3 tablets (600mg) twice daily / 3TC 1 tablet (150mg) twice daily / EFV 1 capsule (600mg) once daily for the duration of 24 weeks
  Interventions: Drug: FZD; Drug: 3TC; Drug: EFV
- FZD 800mg once daily (Experimental): FZD 4 tablets (800mg) once daily / 3TC 2 tablets (150mg) once daily / EFV 1 capsule (600mg) once daily for the duration of 24 weeks
  Interventions: Drug: FZD; Drug: 3TC; Drug: EFV
- FZD 1200mg once daily (Experimental): FZD 6 tablets (1200mg) once daily / 3TC 2 tablets (150mg) once daily / EFV 1 capsule (600mg) once daily for the duration of 24 weeks
  Interventions: Drug: FZD; Drug: 3TC; Drug: EFV
- AZT twice daily (Active Comparator): 1 tablet Combivir(AZT 300mg/3TC 150mg) twice daily / EFV 1 capsule (600mg) once daily for the duration of 24 weeks
  Interventions: Drug: 3TC; Drug: EFV; Drug: AZT

INTERVENTIONS:
Drug: FZD
  Other Names: Fozivudine
  Arms: FZD 1200mg once daily; FZD 600mg twice daily; FZD 800mg once daily
Drug: 3TC
  Other Names: Lamivudine
Drug: EFV
  Other Names: Efavirenz
Drug: AZT
  Other Names: Zidovudine
  Arms: AZT twice daily

SUMMARY:
A prospective, multicenter, open, randomized Phase 2a trial to confirm a sustained virological suppression defined as HIV-RNA <50 copies/ml of 3 different doses of Fozivudine in context to a standard Zidovudine based antiretroviral therapy regimen after 24 weeks of treatment in ART naïve, non subtype B HIV-1 infected individuals from Tanzania and Ivory Coast.

DETAILED DESCRIPTION:
The study will evaluate four different oral 1st line antiretroviral regimens: three study arms will contain different doses of Fozivudine (FZD) plus Lamivudine (3TC) in a twice daily or once daily application plus once daily Efavirenz. The 4th study arm will contain standard Zidovudine (AZT)/Lamivudine (3TC) twice daily in a fixed dose combination plus once daily Efavirenz. The treatment duration will be 24 weeks.

In a pharmacokinetic Sub-Study Pharmacokinetic (PK) characteristics will be determined under controlled conditions in a sub population to evaluate PK values of the study drugs.

Primary Objective

The primary objective is to confirm a sustained virological suppression (HIV RNA <50 copies/ml) after 24 weeks of treatment between three different doses of Fozivudine (FZD) based antiretroviral 1st line treatment regimen in context to a standard Zidovudine (ZDV) based treatment regimen in non subtype B HIV-1 infected individuals from Africa.

Secondary Objectives

1. HIV-RNA log10 reduction of HIV-RNA at 2, 4 and 8 weeks of treatment between different arms
2. Virological response (HIV RNA <50 copies/ml) at 8 and 12 weeks of treatment between different arms
3. Virological response (HIV RNA <400 copies/ml) at 8, 12 and 24 weeks of treatment between different arms
4. Immunologic response: variation in CD4 lymphocytes between different arms
5. Drug toxicity, particularly anaemia, neutropenia and gastrointestinal adverse events
6. Resistance pattern for in patients with virological failure
7. Clinical trial capacity building of African study sites within the FATI network
8. Establishment of a Fozivudine Drug developing consortium (NET) including members of pharmaceutical manufacturers in Asia, Africa and Europe.
9. Development and piloting of a capacity development monitoring and evaluation framework

Pharmacological Objectives

1. Pharmacokinetic assessments after the first intake of study drugs in a subset of study participants (Pharmacokinetic sub study)
2. Pharmacokinetic assessments at steady state after four weeks of study drugs in a subset of study participants (Pharmacokinetic sub study)

Study Population and Study Duration

A total of 120 ART naive HIV-1 infected individuals with the indication to start antiretroviral treatment according to WHO and country guidelines will be enrolled at two study sites in Côte d'Ivoire and Tanzania. Each of the two sites will enroll 60 participants (15 participants per arm). For the PK Sub-Study 6 participants per study arm (total 24 participants will be included.

A minimum of 30% gender representation (female or male) participants will be requested per site. Recruitment, screening and enrollment of study participants are expected to be completed after 9 months. Patient treatment is 24 weeks. So patient related study procedures will take 15 months.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years of age.
2. Provide written or thump printed informed consent prior to all trial-related procedures
3. HIV-1 positive with an indication to start antiretroviral therapy (ART) according to WHO and/or country guidelines
4. ART naïve, including no history of antiretroviral medication during PMTCT or PEP
5. Patient agrees not to take any concomitant medication during the trial without informing the investigator. Traditional medicines should be specified with concomitant medications.
6. Availability throughout the study
7. Female patients of childbearing potential must have a negative pregnancy test and agree to use a highly effective method of birth control throughout participation in the trial and for 10 weeks after last dose (to cover duration of ovulation).
8. Agree to have home visits or active tracing if lost to follow up or any other event justifying a rapid visit of the patient at the clinical trial centre.
9. CD4 count ≥100 cells/μl
10. Hb ≥9.5 g/dl
11. Platelets ≥50,000 cells/mm3
12. Neutrophils ≥500 cells/ mm3
13. Bilirubin <2.5 x uln
14. ALT <2.5 x uln
15. Exclusion of Severe hepatic insufficiency (PT<50%)
16. Creatinine clearance calculated by Cockroft's formula ≥50 ml/min
17. Urine dipstick for protein and blood: negative or trace

Exclusion Criteria:

1. Deficiency in the patient, rendering it difficult, if not impossible, for him/her to take part in the trial or understand the information provided to him/her
2. Presence of an uncontrolled, ongoing, opportunistic infection or of any severe or progressive disease including active TB or any other justified reason which in the opinion of the investigator could significantly inhibit study procedures. This includes any clinical signs possibly associated with any WHO stage 3 or 4, with still unconfirmed diagnosis such as fever, weight loss, diarrhoea or unexplained cough.
3. HIV-2 infection
4. Pregnancy or lactating mother
5. Unlikely to comply with protocol as judged by the principal investigator or his designate
6. Use of experimental therapeutic agents within 30 days of study entry.
7. Hepatitis B with positive HBsAg.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-12; Primary Completion 2014-06 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with plasma HIV RNA < 50 copies/ml | at week 24

SECONDARY OUTCOMES:
Proportion of patients with plasma HIV RNA <50 copies/ml | at week 8 and 12
Proportion of patients with plasma HIV RNA < 400 copies/ml | at week 8, 12 and 24
Mean HIV log10 reduction compared to baseline | at week 2, 4 and 8
Variation of circulating total lymphocyte count | up to week 24
Variation of circulating CD4+ lymphocyte count | up to week 24
Pharmacokinetic parameters (Cmax, AUC, CL/f, CLR, t1/2) before and after the first dose | Day 1
  Various pharmacokinetic parameters (Cmax, AUC, CL/f, CLR, t1/2) will be assessed before the first treatment and during the course of 12 hours after the first treatment.
Pharmacokinetic parameters (Cmax, AUC, CL/f, CLR, t1/2) at steady state | Week 4
  Various pharmacokinetic parameters (Cmax, AUC, CL/f, CLR, t1/2) will be assessed during the course of 12 hours after 4 weeks of treatment.
Proportion of clinical events stage 3 or 4 of WHO HIV classification | up to week 24
Number of participants with Adverse Events as Measure of safety and tolerability | up to week 24
  The number of Adverse Events and also the quality, severity and relatedness to study drug are documented and analysed.
Incidence of resistance mutations after confirmed treatment failure (confirmed HIV RNA > 1000 copies/ml | at week 12 and week 24

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hoelscher, Prof., Study Director — Department for Infectious Diseases and Tropical Medicine, Klinikum of the University of Munich, Leopoldstrasse 5, 80802, Munich, Germany
Locations (2):
- Service des Maladies Infectieuses et Tropicales, CHU de Treichville,, Abidjan, Côte d’Ivoire
- NIMR - Mbeya Medical Research Programme,, Mbeya, Tanzania